CLINICAL TRIAL: NCT01410123
Title: Integrated Stepped Care for Unhealthy Alcohol Use in HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1105008544; U01AA020795 (NIH)
Record Dates: First submitted 2011-07-28; First posted 2011-08-04 (Estimated); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Liver Diseases, Alcoholic; Alcoholism; HIV; Hepatitis C
MeSH Terms: conditions — Liver Diseases, Alcoholic; Alcoholism; Hepatitis C | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment as Usual (TAU) (Other)
  Interventions: Other: Treatment as Usual
- Integrated Stepped Care (ISC) (Other)
  Interventions: Other: Integrated Stepped Care (ISC)

INTERVENTIONS:
Other: Integrated Stepped Care (ISC) — 1. At risk drinking:
     Step 1: Brief negotiated interview (BNI) + booster; Step 2: Motivational Enhancement Therapy; Step 3: Addiction Physician Management + Alcohol pharmacotherapy
  2. Alcohol abuse/dependence:
     Step 1: Addiction Physician Management + Alcohol Pharmacotherapy; Step 2: Motivational Enhancement Therapy; Step 3: Detoxification and aftercare
  3. Moderate Alcohol + Liver Disease:
  Step 1: Brief Negotiated Interview (BNI)+ booster; Step 2: Motivational Enhancement Therapy; Step 3: Addiction physician management + alcohol pharmacotherapy.
  Arms: Integrated Stepped Care (ISC)
Other: Treatment as Usual — The TAU arm will receive a handout with alcohol information embedded within general health-related information (exercise, smoking cessation, and flu vaccination) and standard care as provided by their treating physician. All patients will have access to a NIAAA informational website.
  Arms: Treatment as Usual (TAU)

SUMMARY:
The study is a series of 3 linked randomized clinical trials of 6 month duration, with a total of 12 month follow-up, to evaluate the effect of Integrated Stepped Care on drinking outcomes and HIV biologic markers (including VACS index) in HIV-infected patients with unhealthy alcohol use.

DETAILED DESCRIPTION:
Unhealthy alcohol use threatens the health benefits seen with antiretroviral therapy (ART) for HIV-infected (HIV+) patients. Although research has demonstrated the efficacy of brief interventions, motivational counseling, and medications to treat unhealthy alcohol use in HIV uninfected patients, there is limited research or use of these treatments in HIV+ patients. We have demonstrated that integrated treatment of addiction in HIV clinics is feasible. Stepped care algorithms can facilitate the evaluation of varying intensities of treatments for unhealthy alcohol use. The proposed study will compare onsite Integrated Stepped Care treatment (ISC) to treatment as usual (TAU) in three, linked, 6-month randomized clinical trials in 642 HIV+ patients with unhealthy alcohol use. Screened patients are randomized to ISC or TAU after determining that they meet criteria for either 1) at-risk drinking, 2) alcohol abuse or dependence or 3) moderate alcohol consumption in the presence of liver disease. ISC and TAU are tailored to the drinking category. ISC for at-risk drinkers and those with Moderate Alcohol use and Liver Disease begins with a brief intervention and is stepped up to Motivational Enhancement Therapy (MET) in those who meet predefined failure criteria. ISC for abuse or dependence begins with addiction physician management (APM) including alcohol pharmacotherapy if not contraindicated. APM is stepped up to include MET if predefined failure criteria are met. The study will test the hypothesis that ISC leads to decreased alcohol consumption and improved HIV biomarkers. Data analyses will be conducted on the intention to treat sample.

ELIGIBILITY:
Inclusion Criteria:

1. Be HIV-infected and receiving HIV care at one of the participating medical centers.
2. Meet one of the following criteria for unhealthy alcohol use:

   * At-risk Drinking Study- greater than 14 drinks per week or greater than 4 drinks per occasion in men and greater than 7 drinks per week or greater than 3 drinks per occasion in women and those over 65.
   * Alcohol Abuse or Dependence Study - Meet DSM-IV TR criteria for alcohol abuse or dependence, not in remission.
   * Moderate Alcohol + Liver Disease Study - Report alcohol consumption in the past month, are HCV co-infected, confirmed by HCV viral load or have liver fibrosis - Fib-4 (>1.45). Do not meet criteria for at-risk drinking, alcohol abuse or dependence.
3. Be able to understand English and provide informed consent.

Exclusion Criteria:

1. Be acutely suicidal, or with a psychiatric condition that affects the ability to provide informed consent or participate in counseling interventions (e.g. psychotic, dementia, delusional).
2. Be currently enrolled in formal treatment for alcohol (excluding self-help, e.g. Alcoholics Anonymous)
3. Have medical conditions that would preclude completing or be of harm during the course of the study.
4. Pregnant or nursing women or women who do not agree to use a reliable form of birth control.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 319 (Actual)
Dates: Start 2013-01; Primary Completion 2018-07-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
At risk drinking: Drinks per week | 6 months
Alcohol abuse or dependence: Drinks per week | 6 months
Moderate Alcohol + Liver Disease group: Abstinence. | 6 months

SECONDARY OUTCOMES:
Alcohol consumption by phosphatidylethanol (PEth), an alcohol biomarker | 6 months
Change in biological markers as measured by the VACS index. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: David Fiellin, MD, Principal Investigator — Yale University; Jennifer Edelman, M.D., MHS, Study Director — Yale University
Locations (5):
- United States (5):
  - Washington DC VAMC, Washington D.C., District of Columbia
  - VAMC Atlanta, Atlanta, Georgia
  - New York VAMC - New York Harbor Healthcare System, New York, New York
  - Dallas VA Medical Center, Dallas, Texas
  - VAMC Houston, Houston, Texas

REFERENCES:
- [Background] Edelman EJ, Hansen NB, Cutter CJ, Danton C, Fiellin LE, O'Connor PG, Williams EC, Maisto SA, Bryant KJ, Fiellin DA. Implementation of integrated stepped care for unhealthy alcohol use in HIV clinics. Addict Sci Clin Pract. 2016 Jan 13;11(1):1. doi: 10.1186/s13722-015-0048-z. PMID 26763048
- [Background] Edelman EJ, Maisto SA, Hansen NB, Cutter CJ, Dziura J, Fiellin LE, O'Connor PG, Bedimo R, Gibert C, Marconi VC, Rimland D, Rodriguez-Barradas MC, Simberkoff MS, Justice AC, Bryant KJ, Fiellin DA. The Starting Treatment for Ethanol in Primary care Trials (STEP Trials): Protocol for Three Parallel Multi-Site Stepped Care Effectiveness Studies for Unhealthy Alcohol Use in HIV-Positive Patients. Contemp Clin Trials. 2017 Jan;52:80-90. doi: 10.1016/j.cct.2016.11.008. Epub 2016 Nov 20. PMID 27876616
- [Result] Edelman EJ, Maisto SA, Hansen NB, Cutter CJ, Dziura J, Deng Y, Fiellin LE, O'Connor PG, Bedimo R, Gibert CL, Marconi VC, Rimland D, Rodriguez-Barradas MC, Simberkoff MS, Tate JP, Justice AC, Bryant KJ, Fiellin DA. Integrated stepped alcohol treatment for patients with HIV and liver disease: A randomized trial. J Subst Abuse Treat. 2019 Nov;106:97-106. doi: 10.1016/j.jsat.2019.08.007. Epub 2019 Aug 17. PMID 31540617
- [Result] Edelman EJ, Maisto SA, Hansen NB, Cutter CJ, Dziura J, Deng Y, Fiellin LE, O'Connor PG, Bedimo R, Gibert CL, Marconi VC, Rimland D, Rodriguez-Barradas MC, Simberkoff MS, Tate JP, Justice AC, Bryant KJ, Fiellin DA. Integrated stepped alcohol treatment for patients with HIV and alcohol use disorder: a randomised controlled trial. Lancet HIV. 2019 Aug;6(8):e509-e517. doi: 10.1016/S2352-3018(19)30076-1. Epub 2019 May 17. PMID 31109915
- [Result] Edelman EJ, Maisto SA, Hansen NB, Cutter CJ, Dziura J, Deng Y, Fiellin LE, O'Connor PG, Bedimo R, Gibert CL, Marconi VC, Rimland D, Rodriguez-Barradas MC, Simberkoff MS, Tate JP, Justice AC, Bryant KJ, Fiellin DA. Integrated stepped alcohol treatment for patients with HIV and at-risk alcohol use: a randomized trial. Addict Sci Clin Pract. 2020 Jul 29;15(1):28. doi: 10.1186/s13722-020-00200-y. PMID 32727618
- [Result] Eyawo O, Deng Y, Dziura J, Justice AC, McGinnis K, Tate JP, Rodriguez-Barradas MC, Hansen NB, Maisto SA, Marconi VC, O'Connor PG, Bryant K, Fiellin DA, Edelman EJ. Validating Self-Reported Unhealthy Alcohol Use With Phosphatidylethanol (PEth) Among Patients With HIV. Alcohol Clin Exp Res. 2020 Oct;44(10):2053-2063. doi: 10.1111/acer.14435. Epub 2020 Sep 19. PMID 33460225
- [Result] McGinnis KA, Tate JP, Bryant KJ, Justice AC, O'Connor PG, Rodriguez-Barradas MC, Crystal S, Cutter CJ, Hansen NB, Maisto SA, Marconi VC, Williams EC, Cook RL, Gordon AJ, Gordon KS, Eyawo O, Edelman EJ, Fiellin DA. Change in Alcohol Use Based on Self-Report and a Quantitative Biomarker, Phosphatidylethanol, in People With HIV. AIDS Behav. 2022 Mar;26(3):786-794. doi: 10.1007/s10461-021-03438-y. Epub 2021 Sep 20. PMID 34542779